CLINICAL TRIAL: NCT00520910
Title: Single-Blind Study Determining the Efficacy of Polypodium Leucotomos Extract Supplement in Decreasing UVA Premutagenic and Photoaging Markers
Brief Title: Efficacy of Polypodium Leucotomos Extract Decreasing UVA Premutagenic and Photoaging Markers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Robert S. Kirsner, Professor, University of Miami
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 20070203
Record Dates: First submitted 2007-08-24; First posted 2007-08-27 (Estimated); Results first posted 2019-06-18 (Actual); Last update posted 2019-06-18 (Actual); Status verified 2019-06

CONDITIONS: Aging; Skin Abnormalities
Keywords: Polypodium leucotomos, Ultraviolet Rays, Heliocare, calaguala, anapsos; Skin Aging and Damage
MeSH Terms: conditions — Skin Abnormalities

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Polypodium leucotomos extract (Experimental): Subject is given a 7.5 mg/kg dose of Polypodium leucotomos.
  Interventions: Drug: Polypodium leucotomos
- No intervention (No Intervention): Subject is not given any treatment.

INTERVENTIONS:
Drug: Polypodium leucotomos — Subject is given a 7.5 mg/kg oral dose of Polypodium leucotomos during Baseline visit, and again at 8 hours and 2 hours before the Follow-up visit #2.
  Other Names: Heliocare
  Arms: Polypodium leucotomos extract

SUMMARY:
With this study, the investigators will like to determine if taking a dose of the study medication, called Polypodium leucotomos (PL), prevents some of the changes in the skin caused by the adverse effects of UVA, a type of ultraviolet light.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects,
* 18 years of age or older,
* with Fitzpatrick skin types II and III.

Exclusion Criteria:

* Pregnancy
* Personal history of skin cancer
* History of abnormal photosensitivity
* Smokers
* Patients with history or being exposed to other forms of radiation (other than sunlight)
* History or current exposure to asbestos
* Patients taking any drug that might alter the response of skin to UVR (including, but are not limited to, doxycycline, sulfas, psoralens, and amiodarone)
* Patients unable to undergo skin biopsies
* History of abnormal scarring
* History of adverse reaction to local anesthesia

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2007-08 (Actual); Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian Berman, M.D., Ph.D., Principal Investigator — University of Miami, Department of Dermatology and Cutaneous Surgery
Locations (1):
- University of Miami Skin Research Group Office, Miami, Florida, United States

REFERENCES:
- [Background] Philips N, Smith J, Keller T, Gonzalez S. Predominant effects of Polypodium leucotomos on membrane integrity, lipid peroxidation, and expression of elastin and matrixmetalloproteinase-1 in ultraviolet radiation exposed fibroblasts, and keratinocytes. J Dermatol Sci. 2003 Jun;32(1):1-9. doi: 10.1016/s0923-1811(03)00042-2. PMID 12788523
- [Background] Gombau L, Garcia F, Lahoz A, Fabre M, Roda-Navarro P, Majano P, Alonso-Lebrero JL, Pivel JP, Castell JV, Gomez-Lechon MJ, Gonzalez S. Polypodium leucotomos extract: antioxidant activity and disposition. Toxicol In Vitro. 2006 Jun;20(4):464-71. doi: 10.1016/j.tiv.2005.09.008. Epub 2005 Nov 2. PMID 16263237
- [Background] Alonso-Lebrero JL, Dominguez-Jimenez C, Tejedor R, Brieva A, Pivel JP. Photoprotective properties of a hydrophilic extract of the fern Polypodium leucotomos on human skin cells. J Photochem Photobiol B. 2003 Apr;70(1):31-7. doi: 10.1016/s1011-1344(03)00051-4. PMID 12745244
- [Background] Middelkamp-Hup MA, Pathak MA, Parrado C, Garcia-Caballero T, Rius-Diaz F, Fitzpatrick TB, Gonzalez S. Orally administered Polypodium leucotomos extract decreases psoralen-UVA-induced phototoxicity, pigmentation, and damage of human skin. J Am Acad Dermatol. 2004 Jan;50(1):41-9. doi: 10.1016/s0190-9622(03)02732-4. PMID 14699363
- [Background] Middelkamp-Hup MA, Pathak MA, Parrado C, Goukassian D, Rius-Diaz F, Mihm MC, Fitzpatrick TB, Gonzalez S. Oral Polypodium leucotomos extract decreases ultraviolet-induced damage of human skin. J Am Acad Dermatol. 2004 Dec;51(6):910-8. doi: 10.1016/j.jaad.2004.06.027. PMID 15583582
- [Background] Agar NS, Halliday GM, Barnetson RS, Ananthaswamy HN, Wheeler M, Jones AM. The basal layer in human squamous tumors harbors more UVA than UVB fingerprint mutations: a role for UVA in human skin carcinogenesis. Proc Natl Acad Sci U S A. 2004 Apr 6;101(14):4954-9. doi: 10.1073/pnas.0401141101. Epub 2004 Mar 23. PMID 15041750
- [Background] Berneburg M, Gattermann N, Stege H, Grewe M, Vogelsang K, Ruzicka T, Krutmann J. Chronically ultraviolet-exposed human skin shows a higher mutation frequency of mitochondrial DNA as compared to unexposed skin and the hematopoietic system. Photochem Photobiol. 1997 Aug;66(2):271-5. doi: 10.1111/j.1751-1097.1997.tb08654.x. PMID 9277148
- See also: Skin Research Group Website — http://www.skininvestigation.com

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Polypodium Leucotomos Extract | No Intervention
Started | 5 | 5
Completed | 5 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Polypodium Leucotomos Extract | No Intervention | Total
Number analyzed (Participants) | 5 | 5 | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 5 | 10
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Gender data not collected

OUTCOME MEASURES:

1. Primary Outcome: Change in Common Deletion (CD) Value in DNA of Skin Biopsy Sample
Description: CD is determined by semiquantitative real-time polymerase chain reaction.
Time Frame: baseline, 24 hours
Population: 2 excluded from final data (no detectable baseline common deletion values).
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Polypodium Leucotomos Extract | No Intervention
Number analyzed (Participants) | 5 | 3
percent change | -84 (NA) — Sincere efforts were made to obtain the data from the original PI that left the organization, however, no raw data is available for this outcome. The mean data is available in publication, but the SD was not reported. | 217 (NA) — Sincere efforts were made to obtain the data from the original PI that left the organization, however, no raw data is available for this outcome. The mean data is available in publication, but the SD was not reported.

2. Primary Outcome: 8-oxo-7,8-dihydro-2'-Deoxyguanosine (8-oxo-dG) Quantification in Skin Biopsy Sample Taken From Final Visit
Time Frame: 24 hours
Population: Although data for this outcome measure was collected, however, data are not available. The PI is retired and no longer works in the organization. Sincere efforts were made to obtain the data, however, no data are available for this outcome. Department chair has assume responsibility for this record.
Arm/Group | Polypodium Leucotomos Extract | No Intervention
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 24 hours
Arm/Group | Polypodium Leucotomos Extract | No Intervention
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/5
Other Adverse Events (participants affected / at risk) | 0/5 | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes